CLINICAL TRIAL: NCT00980213
Title: Evaluation of the Cost and Effectiveness in the First-line Treatment of Advanced Renal Cell Cancer With Sunitinib Compared to Interferon-alfa in Finland.
Brief Title: Evaluation of the Cost and Effectiveness Sunitinib Compared to Interferon-Alfa in Finland
Status: Completed | Type: Observational
Sponsor: Pirkko-Liisa Kellokumpu-Lehtinen (Other)
Collaborators: University of Turku (Other); Oulu University Hospital (Other)
Responsible Party: Sponsor-Investigator, Pirkko-Liisa Kellokumpu-Lehtinen, Prof, Tampere University Hospital
Organization: Tampere University Hospital (Other)
Other Study IDs: R09045
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Neoplasms; Renal Cell Carcinoma
Keywords: renal cell cancer; sunitinib; costs; quality of life
MeSH Terms: conditions — Neoplasms; Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sunitinib: advanced renal cell cancer patients treated with sunitinib as first-line therapy
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: sunitinib — sunitinib 50 mg, per os, daily for 4 weeks then 2 weeks pause, duration months

SUMMARY:
Patient receiving sunitinib according the clinician's independent decision as first-line treatment of advanced renal cell carcinoma (RCC) will be asked for informed consent. Treatment with sunitinib will start and end solely on the treating clinicians and the patients independent discretion. Consenting patients will prospectively answer standardized quality of life questionnaires (15D, EQ-5D) during the treatment. Data on health care resource utilisation will be collected prospectively (outpatient visits, hospital stays, concomitant drugs, investigations, sick-leaves, travels). In addition, after treatment failure anti-cancer drugs, hospital stays and date of death will be recorded.

The health economic data during sunitinib treatment and the length of the sunitinib treatment will be compared with the corresponding previously published data collected retrospectively from patients with the same condition treated with IFN-alfa. Stepwise regression analysis will be used to explore whether patient and tumor characteristics explain potential variation in treatment duration and costs that is not explained by the treatment.

Health-related quality of life (HRQoL) data will be presented as descriptive data and compared to age-standardized general population.

At least four major Finnish oncology centers have consented to participate in this study. The inclusion time will be approximately 24 months, and the study time approximately 48 months. Eighty patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Clinically indicated first-line sunitinib treatment for advanced RCC.
* Informed consent obtained.

Exclusion Criteria:

* Unable to complete HRQoL forms.
* Not consenting to collecting register data.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced renal cell cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-09; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incremental cost per incremental time to treatment failure (TTF) in first-line treatment | 1 month

SECONDARY OUTCOMES:
Health related quality of life (HRQoL) | 1 month

CONTACTS AND LOCATIONS:
Locations (5):
- Finland (5):
  - Kuopio University Hospital, Kuopio
  - Oulu Univeristy Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
  - Vaasa Central Hosptital, Vaasa